CLINICAL TRIAL: NCT05900752
Title: A Multi-Strain Probiotic Reduces the Frequency of Diarrhea in IBS-D Patients: A Two-Center, Randomized, Double-Blind, Placebo-controlled Study
Brief Title: A Multi-Strain Probiotic Reduces the Frequency of Diarrhea in IBS-D Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-SM-05-WL-001
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: IBS - Irritable Bowel Syndrome; Diarrhea
Keywords: Probiotics; QiMeiYan
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QiMeiYan Probiotics (Active Comparator): 1.5g/ sachet, containing the following ingredients:
  * Bifidobacterium animalis subsp. lactis V9
  * Lactobacillus casei Zhang
  * Lactobacillus plantarum P-9
  * Lactobacillus plantarum CCFM1143
  * Xylo-oligosaccharide
  * Maltodextrin
  * Resistant Dextrin
  * Blueberry powder
  Interventions: Dietary Supplement: QiMeiYan Probiotics
- Placebo product (Placebo Comparator): 1.5g/sachet, containing the following ingredients:
  * Maltodextrin
  * Blueberry powder
  Interventions: Dietary Supplement: Placebo product

INTERVENTIONS:
Dietary Supplement: QiMeiYan Probiotics — consume one sachet of the assigned product, once a day after meals.
  Arms: QiMeiYan Probiotics
Dietary Supplement: Placebo product — consume one sachet of the assigned product, once a day after meals.
  Arms: Placebo product

SUMMARY:
The goal of this interventional clinical study is to study whether the consumption of QiMeiYan Probiotics in 25-35 young people with Mild irritable bowel syndrome (IBS Score 75 - 175) will reduce the frequency of Diarrhea.

140 eligible participants (70 males and 70 females) will be enrolled in two study sites and randomly assigned to two groups of products QiMeiYan Probiotics and placebo. All participants will consume assigned products once a day after meals and record the critical data such as photo of feces. Three site visits will be arranged and all clinical data will be captured and recorded into CTMS (Clinical Trial Management System) for statistical analysis.

Researchers will compare the two groups to validate if the daily consumption of QiMeiYan Probiotics will reduce the frequency of Diarrhea in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females, age between 25-35, the ratio is 1:1;
* Mild irritable bowel syndrome diagnosed by IBS-SSS, IBS Score 75 - 175;
* Subjects agree not to take any other probiotics during the trial;
* Willing not to participate in other interventional clinical studies during the period of this trial;
* Fully understand the purpose, benefits obtained, possible risks and side effects of the study;
* Willing to comply with all research requirements and procedures;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate.

Exclusion Criteria:

* In the treatment of gastrointestinal symptoms;
* Lactose intolerance;
* Suffering from other organic diseases currently that affect the intestinal function, such as history, colon or rectal cancer resection of gastrointestinal tract, inflammatory bowel disease, diabetes, thyroid function hyperfunction or decline, congenital megacolon, scleroderma, anorexia, etc.;
* Controlling diet, exercising more, or taking medications to control weight or affect appetite in the last 3 months;
* Subjects have any of the following medical history or have been clinically examined to have the following diseases that may affect the evaluation of the test effect: obvious gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases;
* Abuse alcohol or other drugs, supplement or OTC drugs currently or in the past may cause bowel dysfunction or can affect test result evaluation;
* Take drugs frequently that may affect gastrointestinal function or the immune system according to PI's judgment;
* Use laxatives or other substances that promote digestion 2 weeks before the trial;
* Take dairy products or other foods containing prebiotics/bacteria 10 days before the trial.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2023-07-16 (Actual)

PRIMARY OUTCOMES:
Frequency of Diarrhea in IBS-D Patients | baseline day 0, day 28
  Frequency of Diarrhea in IBS-D Patients for the two groups of participants during the study period

SECONDARY OUTCOMES:
Change of Score of IBS-SSS | baseline day 0, day14, day 28
  Change of Score of IBS-SSS for the two groups of participants during the study period. The score of 75-175 is defined as mild severity, 175-300 as middle level severity and >300 as serious level.
Change of Bristol Stool Scale of the feces | baseline day 0, day 7, day 14, day 21, day 28
  Change of Bristol Stool Scale (1-7) of the feces for the two groups of participants during the study period. There are 7 types of feces that matches the look and form of bowel movements indicating potential diarrhea or constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Ruiming Xu, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ai'er Hospital, Shanghai, Shanghai Municipality
  - Meinian Clinical, Chengdu branch, Chengdu, Sichuan

REFERENCES:
- [Background] Merecz K, Hirsa M, Biniszewska O, Fichna J, Tarasiuk A. An overview of 5-HT3 receptor antagonists as a treatment option for irritable bowel syndrome with diarrhea. Expert Opin Pharmacother. 2023 May-Aug;24(10):1189-1198. doi: 10.1080/14656566.2023.2214314. Epub 2023 May 25. PMID 37173833
- [Background] Shaikh OA, Shaikh G, Aftab RM, Baktashi H, Ullah I, Asghar MS. Unconventional but effective: breaking through IBS-D clinical practice guidelines - correspondence. Ann Med Surg (Lond). 2023 Mar 27;85(4):1312-1313. doi: 10.1097/MS9.0000000000000338. eCollection 2023 Apr. PMID 37113818
- [Background] Kim J, Cho K, Kim JS, Jung HC, Kim B, Park MS, Ji GE, Cho JY, Hong KS. Probiotic treatment induced change of inflammation related metabolites in IBS-D patients/double-blind, randomized, placebo-controlled trial. Food Sci Biotechnol. 2019 Dec 23;29(6):837-844. doi: 10.1007/s10068-019-00717-2. eCollection 2020 Jun. PMID 32523793
- [Background] Li Y, Hong G, Yang M, Li G, Jin Y, Xiong H, Qian W, Hou X. Fecal bacteria can predict the efficacy of rifaximin in patients with diarrhea-predominant irritable bowel syndrome. Pharmacol Res. 2020 Sep;159:104936. doi: 10.1016/j.phrs.2020.104936. Epub 2020 May 26. PMID 32470562
- [Background] Ao W, Cheng Y, Chen M, Wei F, Yang G, An Y, Mao F, Zhu X, Mao G. Intrinsic brain abnormalities of irritable bowel syndrome with diarrhea: a preliminary resting-state functional magnetic resonance imaging study. BMC Med Imaging. 2021 Jan 6;21(1):4. doi: 10.1186/s12880-020-00541-9. PMID 33407222
- [Background] Zhang L, Gong M, Tang Y. A commentary on "The efficacy and safety of probiotics in patients with irritable bowel syndrome: Evidence based on 35 randomized controlled trials" (Int J Surg 2020; 75:116-127). Int J Surg. 2020 Apr;76:70. doi: 10.1016/j.ijsu.2020.02.019. Epub 2020 Feb 24. No abstract available. PMID 32105897
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Background] Hellstrom PM. Pathophysiology of the irritable bowel syndrome - Reflections of today. Best Pract Res Clin Gastroenterol. 2019 Jun-Aug;40-41:101620. doi: 10.1016/j.bpg.2019.05.007. Epub 2019 May 24. PMID 31594651
- [Background] Delgado-Herrera L, Lasch K, Zeiher B, Lembo AJ, Drossman DA, Banderas B, Rosa K, Lademacher C, Arbuckle R. Evaluation and performance of a newly developed patient-reported outcome instrument for diarrhea-predominant irritable bowel syndrome in a clinical study population. Therap Adv Gastroenterol. 2017 Sep;10(9):673-687. doi: 10.1177/1756283X17726018. Epub 2017 Aug 24. PMID 28932269
- [Background] Szarka LA, Camilleri M, Burton D, Fox JC, McKinzie S, Stanislav T, Simonson J, Sullivan N, Zinsmeister AR. Efficacy of on-demand asimadoline, a peripheral kappa-opioid agonist, in females with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2007 Nov;5(11):1268-75. doi: 10.1016/j.cgh.2007.07.011. Epub 2007 Sep 27. PMID 17900994
- [Background] Wu H, Zhan K, Rao K, Zheng H, Qin S, Tang X, Huang S. Comparison of five diarrhea-predominant irritable bowel syndrome (IBS-D) rat models in the brain-gut-microbiota axis. Biomed Pharmacother. 2022 May;149:112811. doi: 10.1016/j.biopha.2022.112811. Epub 2022 Mar 15. PMID 35303570
- [Background] Levio S, Cash BD. The place of eluxadoline in the management of irritable bowel syndrome with diarrhea. Therap Adv Gastroenterol. 2017 Sep;10(9):715-725. doi: 10.1177/1756283X17721152. Epub 2017 Jul 24. PMID 28932272
- [Background] Sadrin S, Sennoune S, Gout B, Marque S, Moreau J, Zinoune K, Grillasca JP, Pons O, Maixent JM. A 2-strain mixture of Lactobacillus acidophilus in the treatment of irritable bowel syndrome: A placebo-controlled randomized clinical trial. Dig Liver Dis. 2020 May;52(5):534-540. doi: 10.1016/j.dld.2019.12.009. Epub 2020 Jan 15. PMID 31952938
- [Background] Waller PA, Gopal PK, Leyer GJ, Ouwehand AC, Reifer C, Stewart ME, Miller LE. Dose-response effect of Bifidobacterium lactis HN019 on whole gut transit time and functional gastrointestinal symptoms in adults. Scand J Gastroenterol. 2011 Sep;46(9):1057-64. doi: 10.3109/00365521.2011.584895. Epub 2011 Jun 13. PMID 21663486